CLINICAL TRIAL: NCT05206162
Title: TMS-EEG as a Tool to Study the Neuromodulatory Effects of Theta Burst Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Principal Investigator, Prof. Dr. Kristl Vonck, Prof. Dr. Boon, University Hospital, Ghent
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: EC/2017/0780
Record Dates: First submitted 2022-01-11; First posted 2022-01-25 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-01

CONDITIONS: Cortical Excitability

STUDY DESIGN:
Intervention Model Description: three experimental sessions at randomized order, at least one week apart, in a cross-over design
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- continuous theta burst stimulation (Active Comparator): cTBS over the left motor hotspot, delivered at 80% of resting motor threshold (RMT), according to the Huang et al. protocol, consisting of bursts of stimuli that are presented every 200ms (5Hz), with bursts consisting of 3 stimuli at 50 Hz. A total of 600 pulses are delivered in a continuous train of 40s.
  Interventions: Device: theta burst stimulation
- intermittent theta burst stimulation (Active Comparator): iTBS over the left motor hotspot, delivered at 80% of resting motor threshold (RMT), according to the Huang et al. protocol, consisting of bursts of stimuli that are presented every 200ms (5Hz), with bursts consisting of 3 stimuli at 50 Hz. A total of 600 pulses are delivered in an intermittent train of 190s for iTBS, with repeated cycles of 2s stimulation and 8s pause.
  Interventions: Device: theta burst stimulation
- sham stimulation (Sham Comparator): Sham stimulation over the left motor hotspot, delivered at 80% of resting motor threshold (RMT), according to the Huang et al. protocol, consisting of bursts of stimuli that are presented every 200ms (5Hz), with bursts consisting of 3 stimuli at 50 Hz. A total of 600 pulses are delivered in a continuous train of 40s using a plastic spacer (25mm thickness) between coil and scalp, preventing effective cortical stimulation.
  Interventions: Device: theta burst stimulation

INTERVENTIONS:
Device: theta burst stimulation — TBS over the left motor hotspot, delivered at 80% of resting motor threshold (RMT), according to the Huang et al. protocol, consisting of bursts of stimuli that are presented every 200ms (5Hz), with bursts consisting of 3 stimuli at 50 Hz. A total of 600 pulses are delivered.

SUMMARY:
To assess the effect of continuous (cTBS) and intermittent theta burst stimulation (iTBS) stimulation on motor cortex excitability using TMS-EEG. Based on prior literature, the investigators hypothesized that N100 amplitude would be differently modulated by these two modalities.

DETAILED DESCRIPTION:
Each participant underwent three experimental sessions, at least one week apart in a cross-over design, assessing the effects of a single TBS train over the motor cortex on TMS-evoked potentials measured at the same location and resting-state EEG, immediately before and after the intervention. At each session a different type of TBS was applied (cTBS, iTBS or sham) in a randomized sequence. Subjects were uninformed about the expected effects of each intervention. Sham stimulation was achieved by adding a plastic spacer (25mm thickness) between coil and scalp, preventing effective cortical stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years
* Male
* Right handed subjects
* IQ > 70
* Healthy participants, as determined by history, clinical investigation and investigator's judgment
* No history of central nervous system condition
* No chronic intake of neurotropic drugs
* TMS Safety Screening questionnaire and informed consent signed

Exclusion Criteria:

* Pregnancy, short-term birth wish or childbearing age without adequate birth control
* Intracranial metal hardware (excluding dental filling): surgical clips, shrapnell, electrodes under the stimulation area
* Presence of pacemaker, implantable cardioverter-defibrillator (ICD), permanent medication pumps, cochlear implants or deep brain stimulation (DBS)

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-08-02 (Actual); Primary Completion 2017-11-13 (Actual); Study Completion 2017-11-13 (Actual)

PRIMARY OUTCOMES:
TBS-induced modulation of single-pulse TMS-evoked EEG responses (TEPs) - peak latency/amplitude of TEP components at Cz | measurement takes place immediate before and after TBS stimulation train
TBS-induced modulation of single-pulse TMS-evoked EEG responses (TEPs) - Local Mean Field Power (LMFP) across a region of interest (ROI) | measurement takes place immediate before and after TBS stimulation train
TBS-induced modulation of single-pulse TMS-evoked EEG responses (TEPs) - divergence index (DI) across all EEG channels | measurement takes place immediate before and after TBS stimulation train

SECONDARY OUTCOMES:
TBS-induced modulation of paired-pulse TMS-evoked EEG responses (TEPs) | measurement takes place immediate before and after TBS stimulation train
TBS-induced modulation of resting-state EEG | measurement takes place immediate before and after a single TBS stimulation train

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- [Derived] Carrette S, Vonck K, Klooster D, Raedt R, Carrette E, Delbeke J, Wadman W, Casarotto S, Massimini M, Boon P. Exploration of Theta Burst-Induced Modulation of Transcranial Magnetic Stimulation-Evoked Potentials Over the Motor Cortex. Neuromodulation. 2025 Jan;28(1):123-135. doi: 10.1016/j.neurom.2024.04.007. Epub 2024 Jun 5. PMID 38842956